CLINICAL TRIAL: NCT03667677
Title: Comparison of Tandospirone, Amlodipine and Their Combination in Adults With Hypertension and Anxiety: a Multicentre, Randomized, Double-blind, Double-dummy, Placebo-controlled Trial
Brief Title: Comparison of Tandospirone, Amlodipine and Their Combination in Adults With Hypertension and Anxiety
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Xie Peng, Professor of Neurology, Yongchuan Hospital of Chongqing Medical University, Chongqing Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CES-TAHA
Record Dates: First submitted 2018-09-06; First posted 2018-09-12 (Actual); Last update posted 2018-12-04 (Actual); Status verified 2018-11

CONDITIONS: Hypertension; Anxiety
Keywords: Hypertension; Anxiety; Tandospirone; Amlodipine
MeSH Terms: conditions — Hypertension; Anxiety Disorders | interventions — tandospirone; Amlodipine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1 (Experimental): Tandospirone + Amlodipine
  Interventions: Drug: Tandospirone + Amlodipine
- Group 2 (Experimental): Tandospirone placebo + Amlodipine
  Interventions: Drug: Tandospirone placebo + Amlodipine
- Group 3 (Experimental): Tandospirone + Amlodipine placebo
  Interventions: Drug: Tandospirone + Amlodipine placebo
- Group 4 (Placebo Comparator): Tandospirone placebo + Amlodipine placebo
  Interventions: Drug: Tandospirone placebo + Amlodipine placebo

INTERVENTIONS:
Drug: Tandospirone + Amlodipine — The first group will receive a 30 mg dose of tandospirone one day( a 10 mg dose of tandospirone each time and three times a day) and a 5 mg dose of amlodipine one day(a 5 mg dose of amlodipine and one time a day).
  Arms: Group 1
Drug: Tandospirone placebo + Amlodipine — The second group will receive a 30 mg dose of tandospirone placebo one day( a 10 mg dose of tandospirone placebo each time and three times a day) and a 5 mg dose of amlodipine one day(a 5 mg dose of amlodipine and one time a day).
  Arms: Group 2
Drug: Tandospirone + Amlodipine placebo — The third group will receive a 30 mg dose of tandospirone one day( a 10 mg dose of tandospirone and three times a day) and a 5 mg dose of amlodipine placebo one day(a 5 mg dose of amlodipine placebo and one time a day).
  Arms: Group 3
Drug: Tandospirone placebo + Amlodipine placebo — The fourth group will receive a 30 mg dose of tandospirone placebo one day( a 10 mg dose of tandospirone placebo each time and three times a day) and a 5 mg dose of amlodipine placebo one day(a 5 mg dose of amlodipine placebo and one time a day).
  Arms: Group 4

SUMMARY:
This study compares the antihypertensive effects between different treatment groups including antihypertensive drug, anxiolytic, and both, which provide a new clinical evidence for controlling blood pressure in patients with hypertension and anxiety.

DETAILED DESCRIPTION:
In recent years, many studies have found that elevated blood pressure is associated with anxiety. It has been report that the incidence of hypertension with anxiety is 25%-54%. The studies have confirmed that anxiety can significantly reduce the antihypertensive effect. Therefore, anxiolytics can increase the antihypertensive effect in patients with hypertension and anxiety. However, there is currently no standard treatment for patients with hypertension and anxiety, and few clinical studies have focused on the treatment of these neglected patients. Improvement on hypertension through relieving anxiety and relief of anxiety through lowering hypertension are lack of clinical studies to prove. This study compares the antihypertensive effects between different treatment groups including antihypertensive drug, anxiolytic, and both, which provide a new clinical evidence for controlling blood pressure in patients with hypertension and anxiety.

ELIGIBILITY:
Inclusion Criteria:

1. An age of 60 - 80 years old;
2. Mild or moderate hypertension diagnosed in previous or at screening (office systolic blood pressure ≥ 140 mm Hg and ≤ 180 mm Hg, or diastolic blood pressure ≥ 90 mm Hg and ≤ 110 mm Hg, or both, on three readings on separate days when not taking any blood pressure drugs) ,and the blood pressure still meet the above criteria after the run-in period;
3. A total score ≥ 14 and ≤ 24 on the Hamilton Anxiety Scale (HAMA), except for panic disorder;
4. Informed consent signed.

Exclusion Criteria:

1. Secondary hypertension;
2. Office systolic blood pressure ≥ 180 mm Hg or diastolic blood pressure ≤ 110 mm Hg
3. Hypertension with target organ damage;
4. Cerebral hemorrhage, ischemic cerebral infarction, coronary artery disease, myocardial infarction, second-degree or third-degree atrioventricular block, sick sinus syndrome, atrial fibrillation, left ventricular hypertrophy, cardiac insufficiency (NYHA class Ⅱ-Ⅳ);
5. Diabetes and dyslipidemia;
6. Asthma, chronic obstructive pulmonary disease, bronchiectasis, and respiratory failure;
7. Inflammatory bowel disease, active gastritis, pancreatitis, partial or complete intestinal obstruction, and chronic diarrhea;
8. Acute or chronic hepatitis, hepatic insufficiency (ALT or AST is more than 2 times the upper limit of normal), and renal insufficiency (serum creatinine > 130 umol / L);
9. Uncontrolled thyroid diseases;
10. Severe or unstable central nervous system diseases;
11. Schizophrenia, bipolar disorder, severe intellectual disability, or severe cognitive impairment;
12. Having been diagnosed with alcohol or drug abuse within the past 1 year;
13. Presenting the risk of suicide, self-injury, and hurt others;
14. Having participated in other clinical studies within the past 3 months;
15. Having been treated with anxiolytics, antidepressants, antipsychotics within the past 4 weeks, or have contraindications to the study medications.
16. Breastfeeding, pregnancy, or a pregnancy plan during the study;
17. Other diseases which the responsible clinician judged that a change in current therapy would place the participant at risk.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Estimated)
Dates: Start 2019-02-01 (Estimated); Primary Completion 2020-02-01 (Estimated); Study Completion 2020-07-01 (Estimated)

PRIMARY OUTCOMES:
Office systolic blood pressure and diastolic blood pressure | Change from Baseline Office systolic blood pressure and diastolic blood pressure at 4 weeks and 8 weeks
14-item Hamilton Anxiety Scale(HAMA) | Change from Baseline HAMA score at 4 weeks and 8 weeks
  HAMA-14 are rated on 5 grades ranging from 0(no symptom) to 4 (very severe). The total score ranges from 0 to 56. 29 or more on HAMA means severe anxiety disorders, 21 to 28 on HAMA means obvious anxiety disorders, 14 to 20 on HAMA means anxiety disorders, 8 to 13 on HAMA means suspicious anxiety disorders, 7 or less means no anxiety disorders.

SECONDARY OUTCOMES:
the proportion of patients who met blood pressure control goal( < 140/90mmHg) | Week 8
24-hour ambulatory blood pressure monitoring(ABPM) | Change from Baseline ABPM at 4 weeks and 8 weeks
the proportion of participants with an at least 50% reduction of HAMA score from baseline | Week 8
the proportion of participants showing 7 or less on HAMA | Week 8
20-item Self-Rating Anxiety Scale(SAS) | Change from Baseline SAS score at 4 weeks and 8 weeks
  SAS-20 are rated on 4 grades ranging from 1(a little of the time) to 4(most of the time).The standard score ranges are 25-49 (normal range), 50-59 (mild anxiety), 60-69(moderate anxiety), and 70 or more(severe anxiety).
heart rate variability(HRV) | Change from Baseline HRV at 4 weeks and 8 weeks
17-item Hamilton Depression Rating Scale(HAMD) | Change from Baseline HAMD score at 4 weeks and 8 weeks
  HAMD-17 are rated on 5 grades ranging from 0 (no symptom) to 4 (very severe). 7 or less on HAMD means no depression, 7 to 17 on HAMD means mild depression, 18 to 23 on HAMD means moderate depression, and 24 or more on HAMD means severe depression.
Clinical Global Impression-Improvement(CGI-I) | Change from Baseline CGI-I score at 4 weeks and 8 weeks
Quality of Life Enjoyment and Satisfaction Questionnaire(Q-LES-Q) | Change from Baseline Q-LES-Q score at 4 weeks and 8 weeks
  Q-LES-Q are rated on 5 grades ranging from 1 to 5 points.

CONTACTS AND LOCATIONS:
Locations (7):
- China (7):
  - Beijing Friendship Hospital of Capital Medical University, Beijing, Beijing Municipality
  - Beijing Haidian Section of Peking University Third Hospital, Beijing, Beijing Municipality
  - Xuanwu Hospital of Capital Medical University, Beijing, Beijing Municipality
  - Yongchuan Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Zhongda Hospital of Southeast University, Nanjing, Giangsu
  - Kailuan General Hospital, Tangshan, Hebei
  - the First Affiliated Hospital of Shanxi Medical University, Taiyuan, Shanxi

IPD SHARING:
Plan to Share IPD: No
Any public report on the results of this study will not disclose personal information of the participants.

REFERENCES:
- [Background] Bhattacharya R, Shen C, Sambamoorthi U. Excess risk of chronic physical conditions associated with depression and anxiety. BMC Psychiatry. 2014 Jan 16;14:10. doi: 10.1186/1471-244X-14-10. PMID 24433257
- [Background] Pan Y, Cai W, Cheng Q, Dong W, An T, Yan J. Association between anxiety and hypertension: a systematic review and meta-analysis of epidemiological studies. Neuropsychiatr Dis Treat. 2015 Apr 22;11:1121-30. doi: 10.2147/NDT.S77710. eCollection 2015. PMID 25960656
- [Background] Byrd JB, Brook RD. Anxiety in the "age of hypertension". Curr Hypertens Rep. 2014 Oct;16(10):486. doi: 10.1007/s11906-014-0486-0. PMID 25164965
- [Background] Kretchy IA, Owusu-Daaku FT, Danquah SA. Mental health in hypertension: assessing symptoms of anxiety, depression and stress on anti-hypertensive medication adherence. Int J Ment Health Syst. 2014 Jun 21;8:25. doi: 10.1186/1752-4458-8-25. eCollection 2014. PMID 24987456